CLINICAL TRIAL: NCT04454957
Title: Effectiveness of a Virtual Therapeutic Lifestyle Change Program for Diabetes and Prediabetes
Brief Title: Mastering Diabetes Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Memorial Health System (Other)
Responsible Party: Principal Investigator, David Drozek, Associate Professor, Ohio University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-X-96
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2; PreDiabetes
Keywords: diabetes; prediabetes; glycemia; type 2 diabetes; plant-based diet; nutrition; exercise; obesity / overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Diabetes Mellitus; Motor Activity; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Nonrandomized controlled interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mastering Diabetes (Experimental): Adults (hospital employees, their spouses, and community members) who have been identified as having diabetes or prediabetes based on a health risk assessment, who have chosen to participate in Mastering Diabetes. They may or may not be receiving additional usual care.
  Interventions: Behavioral: Mastering Diabetes
- Usual care (No Intervention): Employees and spouses of the hospital system who are participating in the employee wellness program, who have been identified as having diabetes or prediabetes based on a health risk assessment, who have chosen not to participate in Mastering Diabetes. They may or may not be receiving additional usual care.

INTERVENTIONS:
Behavioral: Mastering Diabetes — Virtual (on-line) lifestyle change program, focused on a plant-based, whole food diet and physical activity.
  Arms: Mastering Diabetes

SUMMARY:
This is a program evaluation that will evaluate the effectiveness of Mastering Diabetes, a therapeutic lifestyle change (TLC) program to control prediabetes and type 2 diabetes.

Lifestyle change, focused on dietary change, physical activity, stress management and control of unhealthy substances has been demonstrated effective in preventing the progression of prediabetes, as well as reversal of diabetes and type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
This will be a nonrandomized controlled study. Participants will self select to be a part of this intervention. The control data will be aggregated matched data from participants in the corporate wellness program at Memorial Health System, who choose not to participate in the intervention.

Study participants will have met the inclusion criteria. Potential participants will be provided with a short summary of this program as a potential activity for their participation, with a link leading to a landing page, which will explain the study in more detail, and will include a link to the consent.

If the potential participant is interested, they can click the link to move to the on line consent. If they agree to the consent, they will be taken to an on line HIPAA release form, which will also need an electronic agreement to be enrolled into the study signified by typing in the participant's name and date of birth.

Once this is completed, an email with an enrollment code and link to Mastering Diabetes will be sent the participant.

Mastering Diabetes Program Description:

The Mastering Diabetes Program is based on the Mastering Diabetes Method, which is based on almost 100 years of evidence based research demonstrating the effectiveness of a low-fat, plant-based, whole-food diet to reverse insulin resistance. Members are provided with a step-by-step online course that educates them how to transition to a low-fat, plant-based, whole-food lifestyle and reduce the overwhelm associated with ineffective pharmaceutical medication and ineffective dietary advice.

The online course provides members with detailed information about the root cause of insulin resistance, the effect of a high-fat diet on increasing insulin resistance, how to achieve excellent blood glucose values in the short-term and in the long-term, what laboratory tests to get to measure progress, an overview of oral diabetes medication and insulin, how to track hour-by-hour decisions for excellent blood glucose control, how to lose weight permanently using a low-fat, plant-based, whole-food diet, how to buy food, where to buy food, how to prepare food easily, the benefits of intermittent fasting for improved insulin sensitivity, how to perform an intermittent fast for excellent results, how to adopt an exercise regimen, how to control your blood glucose before, during, and after exercise, how to change your breakfast, lunch, dinner, and also provides members with a collection of delicious and simple recipes.

The program also provides members with direct access to expert coaches via an online community containing thousands of others living with all forms of diabetes, including type 1 diabetes, type 1.5 diabetes, prediabetes, type 2 diabetes, and gestational diabetes. In addition, members get access to live biweekly Q&A videoconferences in which they can interact with coaches and personalize their experience. The cost of full coaching program is $399 for the first 3 months, then $99 per month thereafter.

Participants, having enrolled in the wellness program, will already, as a part of that study, have agreed to have data collected at baseline and yearly thereafter, including BMI, blood pressure, resting pulse, lipid panel, hemoglobin A1c, health risk assessment survey, absenteeism and health claims data at baseline and yearly thereafter. If not collected within 60 days, a new set of data will be collected to serve as baseline for this study. This is not specific for this study, but is the case for any new program activity that a participant in the corporate wellness study begins.

Specifically for this study the health risk assessment data collection (including lab analysis) will also be repeated at 12 weeks. The lab work is accomplished at any MHS lab facility, according to current medical system standards.

Participant health claims data will also be evaluated, beginning with the prior year's data, if available from MHS Human Resources, being utilized as a baseline, and followed for the subsequent years of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years at enrollment
* Has a diagnosis of diabetes or prediabetes or a HbA1c of 5.7 or higher.
* Are able to participate in physical activity.
* Are willing to use a smartphone or computer to access the online education modules and online community, and have reliable daily Internet access with a device with a webcam
* Have an email account and an Internet connection at home
* Are able to purchase and transport fresh produce from a local grocery store to their house on a weekly basis
* Are able to prepare food in their house or get help preparing food in their house following recipes and meal examples provided in the online course
* Are open-minded about eating a plant-based diet, performing periodic intermittent fasting (16-24 hours, once a week),
* Are willing to increase movement of their body 5-6 days per week
* Are willing to participate in an online community for support and coaching
* Are willing to participate in biweekly videoconferencing for support and coaching
* Are willing to be courteous and respectful to others in the online community

Exclusion Criteria:

* Has been told by a medical provider to not participate in physical activity.
* Has a medical condition that prevents walking at least a mile a day.
* Deemed unsuitable to exercise by Dr. Drozek or other members of the wellness team.
* Has a diagnosis of dementia.
* Is pregnant or planning to become pregnant during the program
* Does not speak or understand English
* Advanced renal disease (stage 4 or 5) with or without hemodialysis
* Congestive heart failure
* Has inflammatory bowel disease (Crohns disease, ulcerative colitis)
* Is fed by a feeding tube
* Is taking Coumadin or warfarin
* Inability to use email, a smartphone, or the Internet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c | up to 20 years
  glycosylated hemoglobin measured from venous blood
BMI | up to 20 years
  Body mass index calculated from height and weight
Healthcare expenditures | up to 20 years
  Monetary amount spent for healthcare

SECONDARY OUTCOMES:
Total cholesterol | baseline, 12 weeks, 1 yearly, then yearly for up to 20 years
  Measured from a lipid panel done on venous blood
Low density lipoprotein cholesterol | baseline, 12 weeks, 1 yearly, then yearly for up to 20 years
  Calculated from a lipid panel done on venous blood
High density lipoprotein cholesterol | baseline, 12 weeks, 1 yearly, then yearly for up to 20 years
  Measured from a lipid panel done on venous blood
Triglyceride | baseline, 12 weeks, 1 yearly, then yearly for up to 20 years
  Measured from a lipid panel done on venous blood
Exercise level | baseline, 12 weeks, 1 yearly, then yearly for up to 20 years
  Amount of time spent per week in moderate to vigorous physical activity
Dietary Recall | baseline, 12 weeks, 1 yearly, then yearly for up to 20 years
  Daily or weekly average of foods consumed during the last 7 days
Patient Health Questionnaire | baseline, 12 weeks, 1 yearly, then yearly for up to 20 years
  mood screening questions; two for anxiety
Patient Health Questionnaire | baseline, 12 weeks, 1 yearly, then yearly for up to 20 years
  mood screening questions; two for depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Retrospective Evaluation of an Online Diabetes Health Coaching Program: A Pilot Study — https://pubmed.ncbi.nlm.nih.gov/34366745/